CLINICAL TRIAL: NCT00478088
Title: A Pivotal, Multi-Center, Randomized, Controlled Trial Evaluating The Safety and Effectiveness of The NeoDisc™ Versus Instrumented Anterior Cervical Discectomy and Fusion (ACDF) in Subjects With Single-Level Cervical Disc Disease
Brief Title: Evaluating The Safety and Effectiveness of The NeoDisc™ Versus ACDF in Subjects With Single-Level Cervical Disc Disease
Acronym: NeoDisc™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NUVA-ND-0501
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2012-05

CONDITIONS: Cervical Disc Degenerative Disorder
Keywords: Single Level; Cervical Disc Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): NeoDisc
  Interventions: Device: NeoDisc
- 2 (Active Comparator): ACDF
  Interventions: Device: Instrumented Anterior Cervical Discectomy and Fusion (ACDF)

INTERVENTIONS:
Device: NeoDisc — The NeoDisc is an artificial cervical intervertebral disc replacement intended for clinical use following a discectomy.
  Arms: 1
Device: Instrumented Anterior Cervical Discectomy and Fusion (ACDF) — Surgical removal of the cervical disc, decompression, and anterior implantation of allograft bone with a cervical plate.
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the NeoDisc compared to anterior cervical discectomy and fusion (ACDF) for the treatment of single-level cervical disc disease, by demonstrating non-inferior comparative results at the 24 month follow-up period pertaining to (1) improvement in the Neck Disability Index (NDI) score, (2) revision/reoperation/removal rate, (3) complication rate, and (4) maintenance or improvement in neurologic status.

DETAILED DESCRIPTION:
The NeoDisc is an artificial cervical intervertebral disc replacement intended for clinical use following a discectomy. Implantation of the device will result in artificial replacement of a pathologically damaged or surgically removed cervical disc. Use of the device also obviates the need to harvest bone graft from the patient's iliac crest, a common and painful part of current surgical techniques.

The NeoDisc is indicated for cervical spinal arthroplasty in skeletally mature subjects with symptomatic cervical disc disease at one level from C3 to C7. Symptomatic cervical disc disease is defined as image-confirmed herniated disc, spondylosis, and/or loss of disc height, with functional neurological deficit (i.e., exhibits at least one sign associated with cervical level to be treated, including abnormal reflex, decreased motor strength, abnormal dermatome sensitivity, or pain in a dermatomal distribution).

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age (inclusive and skeletally mature)
* Diagnosis of symptomatic cervical disc disease, defined as image- confirmed pathology: herniated disc, spondylosis, and/or loss of disc height. Spondylosis is defined as MRI or CT-confirmed disc dessication, loss of disc height, bridging osteophytes, and/or uncovertebral arthrosis. Loss of disc height is specified as a measurement of at least 25% less than an adjacent nonsymptomatic level, but with a minimum of 1mm height remaining.
* Functional neurological deficit (i.e., exhibits at least one sign associated with cervical level to be treated, including abnormal reflex, decreased motor strength, abnormal dermatome sensitivity, or pain in a dermatomal distribution)
* Symptomatic level is C3-4, C4-5, C5-6 or C6-7 (one level)
* Preop NDI ≥30 points
* Unresponsive to conservative treatment for ≥6 wks, or exhibits progressive symptoms or signs of nerve root or spinal cord compression in the face of conservative treatment
* Not pregnant, nor interested in becoming pregnant within the follow-up period of the study
* Willing and able to comply with the requirements defined in the protocol for the duration of the study
* Signed and dated Informed Consent

Exclusion Criteria:

* Prior cervical fusion surgery at the operative level
* Prior cervical laminectomy at the operative level (prior cervical laminotomy need not be excluded)
* Prior cervical complete facetectomy at the operative level
* Requiring surgical treatment that would leave the patient with a postoperative deficiency of the posterior elements
* Radiographic signs of significant instability at operative level (greater than 3mm translation, > 11 degrees rotation different from adjacent level)
* Bridging osteophytes or motion < 2 degrees
* Radiographic confirmation of significant facet joint disease or degeneration
* Chronic neck or arm pain of unknown etiology
* Clinically significant symptomatic myelopathy (e.g., those with signal changes in the spinal cord on preoperative T2-weighted MRI)
* Cervical fracture, anatomic anomaly, or deformity (e.g. ankylosing spondylitis, scoliosis) at the levels to which the prosthesis will be attached
* Severe spondylolisthesis (>grade 1)
* Endocrine disorders or connective tissue diseases
* Rheumatoid arthritis or other autoimmune disease
* Progressive neuromuscular disease, e.g., muscular dystrophy, multiple sclerosis
* Chronic steroid users
* Taking any medications or drugs that are known to potentially interfere with the bone metabolism or soft tissue healing, which may include (but is not limited to) the following: inhaled glucocorticoids for asthma, corticosteroids, thyroid hormones, blood thinners (heparin, warfarin), gonadotropin-releasing hormone agonists for prostate cancer treatment, contraceptive medroxyprogesterone, lithium for bi-polar disorder treatment, anticonvulsants, aluminum-containing antacids, tetracycline
* Osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated (DEXA T-score less than or equal to -2.5; DEXA necessary only if patient exhibits risk factors for low bone mass as quantified in DEXA screening questionnaire).
* Diabetes mellitus requiring insulin management
* Presence of metastases or active spinal tumor malignancy
* Body Mass Index (BMI) > 40
* Active local or systemic infection, including AIDS, hepatitis
* Having been enrolled in another investigational device study within the last 90 days
* Having had another cervical device implanted that would interfere with the surgical approach, study or control device, or follow-up evaluations.
* Demonstrates signs of nonorganic behavior, such as Waddell's signs
* History of substance abuse
* Involved in spinal litigation
* Mentally incompetent
* Incarcerated

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 488 (Actual)
Dates: Start 2006-09; Primary Completion 2010-08 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Improve in NDI by ≥ 15 pnts at 24 mo compared to Baseline; No device failures requiring revision, re-op or removal; No major complications,i.e.,vascular or neurological injury; Maintenance or improvement of neurologic status | August 2010

SECONDARY OUTCOMES:
ROM; Fusion/migration of device; SF-36 imp of ≥15% at 24 months comp to Baseline; VAS imp of > 20 mm at 24 months comp to Baseline; Disc ht from lateral x-ray showing maintenance or imp from Baseline at 24 | August 2010

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kitchel, MD, Principal Investigator — Medical Monitor
Locations (22):
- United States (22):
  - San Diego Center for Spinal Disorders, La Jolla, California
  - Diagnostic and Interventional Surgical Center, Marina del Rey, California
  - The Spine Institute, Santa Monica, California
  - Spine Colorado / Durango Orthopedic Associates, Durango, Colorado
  - Rocky Mountain Spine Arthroplasty (RMA Ortho), Loveland, Colorado
  - Florida Spine Specialists, Fort Lauderdale, Florida
  - Florida Research Network, LLC, Gainesville, Florida
  - Lyerly Baptist, Jacksonville, Florida
  - Optim Healthcare, Savannah, Georgia
  - OAD Orthopaedics, Warrenville, Illinois
  - OrthoIndy, Indianapolis, Indiana
  - Spine Midwest, Inc, Jefferson City, Missouri
  - Western Regional Spine Center for Brain and Spine Surgery, Las Vegas, Nevada
  - Coastal Spine, Mount Laurel, New Jersey
  - Capital Neurosurgery, Raleigh, North Carolina
  - Center for Advanced Orthopaedics/Adena Health Pavillon, Chillicothe, Ohio
  - Neurological Associates, Columbus, Ohio
  - Central Ohio Neurological Surgeons, Westerville, Ohio
  - Orthopedic Spine Associates, Eugene, Oregon
  - Southern Oregon Orthopedics, Medford, Oregon
  - Central Texas Spine Institute, Austin, Texas
  - Salt Lake Orthopaedic Clinic, Salt Lake City, Utah